CLINICAL TRIAL: NCT02770521
Title: A Study to Evaluate the Safety and Tolerability of Subcutaneous Treprostinil and Pharmacokinetics of a Novel LY900014 Formulation in Healthy Japanese Subjects
Brief Title: A Study of Treprostinil and a New Formulation of LY900014 in Healthy Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 16071; I8B-JE-ITRK (Other: Eli Lilly and Company)
Record Dates: First submitted 2016-05-11; First posted 2016-05-12 (Estimated); Results first posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2016-07

CONDITIONS: Healthy
MeSH Terms: interventions — treprostinil; Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treprostinil (Part A) (Experimental): Treprostinil administered as a single subcutaneous (SC) bolus injection.
  Interventions: Drug: Treprostinil
- Placebo (Part A) (Placebo Comparator): Placebo administered as a single SC bolus injection.
  Interventions: Drug: Placebo
- LY900014 (Part B) (Experimental): LY900014 (test) administered as a single SC bolus injection.
  Interventions: Drug: LY900014
- Insulin Lispro (Part B) (Active Comparator): Insulin lispro (reference) administered as a single SC bolus injection.
  Interventions: Drug: Insulin Lispro

INTERVENTIONS:
Drug: Treprostinil — Administered SC.
  Arms: Treprostinil (Part A)
Drug: Placebo — Administered SC.
  Arms: Placebo (Part A)
Drug: LY900014 — Administered SC.
  Other Names: Ultra-Rapid Lispro
  Arms: LY900014 (Part B)
Drug: Insulin Lispro — Administered SC.
  Arms: Insulin Lispro (Part B)

SUMMARY:
The aims of this study are to evaluate:

* The safety and tolerability of a single dose of treprostinil given subcutaneously (as an injection just under the skin)
* The pharmacokinetic profile (how the body absorbs, breaks down, and gets rid of) of a single subcutaneous dose of a new LY900014 formulation in healthy Japanese participants.

The study has two parts. Participants may only enroll in one part.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy Japanese
* Body mass index (BMI) 18.5 - 25 kilograms per square meter (kg/m²)
* Fasting plasma glucose ≥71 milligrams per deciliter (mg/dL) (3.9 millimoles per liter [mmol/L]) and <108 mg/dL (6.0 mmol/L) (Part B only)
* Have normal blood pressure, pulse rate, electrocardiogram (ECG), blood and urine laboratory test results that are acceptable for the study

Exclusion Criteria:

* Are currently enrolled in a clinical trial involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study
* Have participated in a clinical trial involving an investigational product within the 30 days before study entry.
* Have previously completed or withdrawn from this study or any other study investigating treprostinil or LY900014, and have previously received the investigational product
* Have or used to have health problems or laboratory test results or ECG readings that, in the opinion of the doctor, could make it unsafe to participate, or could interfere with understanding the results of the study

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-05; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study had two parts: Part A was a two-period crossover. Part B was a three-period crossover with dose escalation. Healthy Japanese participants were eligible to enroll in one part. One randomized participant discontinued prior to study completion and was replaced. The replacement adopted the original participant's randomization scheme.
Groups:
- Placebo/Treprostinil (Part A): Placebo given subcutaneously (SC) once in first study period. 1,000 nanograms (ng) of treprostinil given SC once in second study period. There was a minimum three day washout between doses.
- Treprostinil/Placebo (Part A): 1,000 ng of treprostinil given SC once in first study period. Matching placebo given SC once in second study period. There was a minimum three day washout between doses.
- 15 U Insulin Lispro/15 U LY900014/30 U LY900014 (Part B): 15 units (U) insulin lispro given SC once in first study period. 15 U LY900014 given SC once in second study period. 30 U LY900014 given SC once in third study period. There was a minimum three day washout between doses.
- 7.5 U LY900014/15 U Insulin Lispro/30 U LY900014 (Part B): 7.5 U LY900014 given SC once in first study period. 15 U insulin lispro given SC once in second study period. 30 U LY900014 given SC once in third study period. There was a minimum three day washout between doses.
- 7.5 U LY900014/15 U LY900014/15 U Insulin Lispro (Part B): 7.5 U LY900014 given SC once in first study period. 15 U LY900014 given SC once in second study period. 15 U insulin lispro given SC once in third study period. There was a minimum three day washout between doses.
- 7.5 U LY900014/15 U LY900014/30 U LY900014 (Part B): 7.5 U LY900014 given SC once in first study period. 15 U LY900014 given SC once in second study period. 30 U LY900014 given SC once in third study period. There was a minimum three day washout between doses.
Period: Period One
Arm/Group | Placebo/Treprostinil (Part A) | Treprostinil/Placebo (Part A) | 15 U Insulin Lispro/15 U LY900014/30 U LY900014 (Part B) | 7.5 U LY900014/15 U Insulin Lispro/30 U LY900014 (Part B) | 7.5 U LY900014/15 U LY900014/15 U Insulin Lispro (Part B) | 7.5 U LY900014/15 U LY900014/30 U LY900014 (Part B)
Started | 4 | 4 | 2 | 2 | 2 | 9
Received Study Drug | 4 | 4 | 2 | 2 | 2 | 9
Completed | 4 | 4 | 2 | 2 | 2 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period Two
Arm/Group | Placebo/Treprostinil (Part A) | Treprostinil/Placebo (Part A) | 15 U Insulin Lispro/15 U LY900014/30 U LY900014 (Part B) | 7.5 U LY900014/15 U Insulin Lispro/30 U LY900014 (Part B) | 7.5 U LY900014/15 U LY900014/15 U Insulin Lispro (Part B) | 7.5 U LY900014/15 U LY900014/30 U LY900014 (Part B)
Started | 4 | 4 | 2 | 2 | 2 | 9
Received Study Drug | 4 | 4 | 2 | 2 | 2 | 9
Completed | 4 | 4 | 2 | 2 | 2 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period Three
Arm/Group | Placebo/Treprostinil (Part A) | Treprostinil/Placebo (Part A) | 15 U Insulin Lispro/15 U LY900014/30 U LY900014 (Part B) | 7.5 U LY900014/15 U Insulin Lispro/30 U LY900014 (Part B) | 7.5 U LY900014/15 U LY900014/15 U Insulin Lispro (Part B) | 7.5 U LY900014/15 U LY900014/30 U LY900014 (Part B)
Started | 0 (Not applicable. Part A only had two periods.) | 0 (Not applicable. Part A only had two periods.) | 2 | 2 | 2 | 9
Received Study Drug | 0 | 0 | 2 | 2 | 2 | 9
Completed | 0 | 0 | 2 | 2 | 2 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Treprostinil or Placebo (Part A): Participants received either 1000 ng of treprostinil or matching placebo as a SC injection once in each of two study periods.
- LY900014 or Insulin Lispro (Part B): Participants received each of three doses of LY900014 (7.5 U, 15 U, 30 U) or 15 U of insulin lispro as a SC injection once in each of three study periods.
- Total: Total of all reporting groups
Arm/Group | Treprostinil or Placebo (Part A) | LY900014 or Insulin Lispro (Part B) | Total
Number analyzed (Participants) | 8 | 15 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.3 (4.4) | 26.1 (5.4) | 26.2 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 15 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 15 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 15 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 8 | 15 | 23
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per meter squared (kg/m²)] | 22.57 (2.00) | 21.93 (2.19) | 22.15 (2.10)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, are reported in the Adverse Events module.
Time Frame: Part A: Baseline through Study Completion (up to 14 Days after Last Dose)
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: participants
Groups:
- Placebo (Part A): Placebo given subcutaneously (SC) once in one of two study periods. There was a minimum three day washout between doses.
- Treprostinil (Part A): 1,000 ng of treprostinil given SC once in one of two study periods. There was a minimum three day washout between doses.
- 15 U Insulin Lispro (Part B): 15 units (U) insulin lispro given SC once in up to one of three study periods. There was a minimum three day washout between doses.
- 7.5 U LY900014 (Part B): 7.5 U LY900014 given SC once in up to one of three study periods. There was a minimum three day washout between doses.
- 15 U LY900014 (Part B): 15 U LY900014 given SC once in up to one of three study periods. There was a minimum three day washout between doses.
- 30 U LY900014 (Part B): 30 ULY900014 given SC once in up to one of three study periods. There was a minimum three day washout between doses.
Arm/Group | Placebo (Part A) | Treprostinil (Part A) | 15 U Insulin Lispro (Part B) | 7.5 U LY900014 (Part B) | 15 U LY900014 (Part B) | 30 U LY900014 (Part B)
Number analyzed (Participants) | 8 | 8 | 6 | 13 | 13 | 13
participants | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Pharmacokinetics (PK): Insulin Lispro Maximum Concentration (Cmax) (Part B)
Description: PK: Insulin Lispro Cmax (Part B)
Time Frame: Predose, 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, 55, 60, 70, 90, 120, 150, 180, 240, 300, 360, and 420 Minutes Postdose
Population: All participants who received at least one dose of study drug LY900014 in Part B and had evaluable pharmacokinetic data. Per protocol, PK in Part B was not analyzed for 15 U Insulin Lispro (Humalog). This arm was included for only safety analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomoles/liter (pmol/L)
Groups:
- 30 U LY900014 (Part B): 30 U LY900014 given SC once in up to one of three study periods. There was a minimum three day washout between doses.
Arm/Group | 7.5 U LY900014 (Part B) | 15 U LY900014 (Part B) | 30 U LY900014 (Part B)
Number analyzed (Participants) | 13 | 13 | 13
picomoles/liter (pmol/L) | 582 (42) | 956 (41) | 2170 (30)

3. Primary Outcome: PK: Insulin Lispro Area Under the Concentration-Time Curve From Time Zero to 30 Minutes (AUC[0-30min]) (Part B)
Description: PK: Insulin Lispro AUC(0-30min) (Part B)
Time Frame: Predose, 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, 55, 60, 70, 90, 120, 150, 180, 240, 300, 360, and 420 Minutes Postdose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol*hour/L (pmol*hr/L)
Arm/Group | 7.5 U LY900014 (Part B) | 15 U LY900014 (Part B) | 30 U LY900014 (Part B)
Number analyzed (Participants) | 13 | 13 | 13
pmol*hour/L (pmol*hr/L) | 174 (57) | 273 (51) | 585 (31)

4. Secondary Outcome: PK: Treprostinil Time to Maximum Concentration (Tmax) (Part A)
Description: PK: Treprostinil Tmax (Part A)
Time Frame: 15, 30, 60 and 120 Minutes Postdose
Population: All participants in Part A who received study drug and had evaluable pharmacokinetic data.
Measure: Median (Full Range); unit: hours
Groups:
- Treprostinil (Part A): 1,000 ng treprostinil administered as a single subcutaneous (SC) injection in one of two study periods.
Arm/Group | Treprostinil (Part A)
Number analyzed (Participants) | 8
hours | 0.25 [0.25 to 0.50]

5. Secondary Outcome: PK: Maximum Concentration (Cmax) of Treprostinil (Part A)
Description: PK: Cmax of Treprostinil (Part A)
Time Frame: 15, 30, 60 and 120 Minutes Postdose
Population: All participants in Part A who received study drug and had evaluable pharmacokinetic data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/milliliter (mL)
Arm/Group | Treprostinil (Part A)
Number analyzed (Participants) | 8
ng/milliliter (mL) | 0.0271 (36)

ADVERSE EVENTS:
Time Frame: Baseline through Study Completion (up to 14 Days after Last Dose)
Description: All participants who received at least one dose of study drug.
Arm/Group | Placebo (Part A) | Treprostinil (Part A) | 15 U Insulin Lispro (Part B) | 7.5 U LY900014 (Part B) | 15 U LY900014 (Part B) | 30 U LY900014 (Part B)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/6 | 0/13 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/6 | 0/13 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/8 | 5/8 | 3/6 | 7/13 | 7/13 | 2/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Part A) (N=8) | Treprostinil (Part A) (N=8) | 15 U Insulin Lispro (Part B) (N=6) | 7.5 U LY900014 (Part B) (N=13) | 15 U LY900014 (Part B) (N=13) | 30 U LY900014 (Part B) (N=13)
Infusion site phlebitis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Injection site erythema (General disorders) | 0 (0) | 5 (5) | 3 (3) | 7 (7) | 6 (6) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days